CLINICAL TRIAL: NCT01577784
Title: A Phase II, Opened, Not Controlled and Multicentric Clinical Trial of Pazopanib in Monotherapy to Determine Efficiency and Safety in Second-line of Treatment in Patients With Carcinoma of Advanced Renal Cells That Have Progressed or Have Not Tolerated the First Line of Treatment With Tyrosine Kinase Inhibitor
Brief Title: Pazopanib in Second-line Therapy in Renal Cell Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Associació per a la Recerca Oncologica, Spain (Other)
Collaborators: Trial Form Support S.L. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APRO02-2011
Record Dates: First submitted 2012-04-10; First posted 2012-04-16 (Estimated); Last update posted 2014-03-12 (Estimated); Status verified 2014-03

CONDITIONS: Metastatic Renal Cell Carcinoma
Keywords: Advanced renal cell carcinoma; second-line treatment with pazopanib; first line of treatment with a Tyrosine Kinase Inhibitor
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — pazopanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pazopanib (Experimental): 800 mg / day of pazopanib in monotherapy
  Interventions: Drug: Pazopanib

INTERVENTIONS:
Drug: Pazopanib — 800 mg / day of pazopanib in monotherapy.
  Other Names: Pazopanib (GW786034; Votrient®)

SUMMARY:
The principal aim of the study is to determine the objective response rate that offers the second-line treatment with pazopanib in patients with carcinoma of advanced renal cells that have progressed or that have not tolerated the first line of treatment with a Tyrosine Kinase Inhibitor. The secondary aims are to determine the overall survival and the treatment safety profile for these patients in second-line treatment with pazopanib. The exploratory aim is to determine the correlation between biomarkers in patient blood and tumor samples, and the clinical results obtained with pazopanib.

DETAILED DESCRIPTION:
Patients who progress or do not tolerate a first-line treatment with a Tyrosine Kinase Inhibitor will be included consecutively in the study. All patients will receive the same treatment regimen consisting of 800 mg / day of pazopanib in monotherapy.

All patients will receive treatment until there is evidence of progression, evidence of unacceptable toxicity, not compliance, investigator clinical decision or consent withdrawal by the patient.

After treatment, the patient will enter to the follow-up period. During this period the investigator will collect information from subsequent administered treatments and survival of all patients, regardless of the reason for withdrawal, every 8 weeks until the scheduled end of follow-up period, according to protocol. At 30 days after treatment completion, the first follow up visit will be scheduled to assess the possible occurrence of late toxicity. In those patients who complete treatment prior to objectify progression, information about the progression of the disease will be collected.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Inform Consent
2. Age ≥ 18
3. Histologically confirmed diagnosis of clear cell renal carcinoma metastatic or locally recurrent unresectable.
4. Patients must have received only a first-line treatment with a Tyrosine Kinase Inhibitor. Patients must have progressed during treatment or within three months after stopping treatment with these agents. Patients who discontinued treatment with a Tyrosine Kinase Inhibitor for unacceptable toxicity are also eligible for the study.
5. Patients must have been previously treated by nephrectomy with removal of the primary tumor, except that there is a contraindication (eg liver I extensive bone metastatic disease or primary tumor smaller than 5 cm).
6. Patients with ECOG PS 0 or 1.
7. To be included in the study, the renal tumor should be classified in a group of low or intermediate risk according to the Motzer classification.
8. Eligibility criteria under RECIST v.1.1
9. Adequate hematologic function:

   Absolute neutrophil count ≥ 1.5 x 109 / L Platelet count ≥ 100 x 109 / L Hemoglobin ≥ 9 g / dL (5.6 mmol / L). Prothrombin time (PT) or international normalized ratio (INR) ≤ 1.2 X ULN. Activated partial thromboplastin time (APTT) ≤ 1.2 X ULN
10. Adequate hepatic function:

    total bilirubin ≤ 1.5 X ULN ALT ≤ 2.5 x ULN
11. Adequate renal function:

    Serum creatinine ≤ or 1.5 mg / dL (133 mol / L). If> 1.5 mg / dL, then the calculated creatinine clearance has to be ≥ 50 mL / min (Appendix 1).

    Urine protein / creatinine ratio <1.
12. Can be included in the study of both fertile and infertile women.

Exclusion Criteria:

1. Previous malignancy. May be included in the study patients with a disease-free interval of 5 years at the time of inclusion in the study and patients with non-melanoma skin carcinoma completely resected or carcinoma in situ treated successfully.
2. Previous treatment with more then one Tyrosine Kinase Inhibitor or more than one previous traditional regime (eg, chemotherapy, immunotherapy or chemo-immunotherapy).
3. Known history or clinical evidence of nervous system metastases or leptomeningeal carcinomatosis, except that metastases in the central nervous system have been previously treated, are asymptomatic and not requiring treatment with corticosteroids or anticonvulsant medication within six months before the first administration of pazopanib.
4. Clinically significant gastrointestinal disorders that may increase the risk of bleeding gastrointestinal.
5. Clinically significant gastrointestinal disorders which may affect the absorption of pazopanib.
6. Presence of uncontrolled infection.
7. ECG QT interval longer than 480 milliseconds, according to the Bazett formula.
8. History of one or more of the following cardiovascular conditions within the last 6 months prior to inclusion:

   Cardiac angioplasty or stent placement Myocardial infarction Unstable angina Surgery or coronary bypass Symptomatic peripheral vascular disease
9. Congestive heart failure Class III or IV, as defined by the New York Heart Association
10. Poorly controlled hypertension (defined as systolic blood pressure ≥ 140 mmHg or diastolic blood pressure ≥ 90 mmHg).
11. History of stroke (including transient ischemic attack), pulmonary embolism or deep vein thrombosis not treated within 6 months.
12. Major surgery or major trauma within 28 days prior to administering the first dose of study and / or presence of any unhealed wound, fracture, or ulcer (not considered major procedures such as venous catheter placement with or without a reservoir).
13. Evidence of bleeding diathesis or active bleeding.
14. Endobronchial lesions known and / or lesions infiltrating major pulmonary vessels.
15. Hemoptysis greater than 2.5 milliliters in the 8 weeks before the first administration of study drug.
16. Any medical condition, psychiatric or any other nature, unstable or severe, which could interfere with patient safety, with the ability to give informed consent or compliance with study procedures.
17. Inability or lack of willingness to discontinue the use of banned drugs listed in in the previous 14 days, or the time equivalent to 5 half-lives (whichever is greater) at baseline and during treatment with pazopanib.
18. Treatment with any of the following antineoplastic therapy: radiation therapy, surgery, tumor embolization, chemotherapy, immunotherapy, biologic therapies, investigational therapies or hormone treatments within 14 days, or the time equivalent to 5 half-lives (whichever is greater), to the administration of the first dose of pazopanib.
19. Any unresolved toxicity from previous cancer therapies> Grade 1 and / or is getting worse in intensity, except for alopecia.
20. Patients who are at risk of hypersensitivity to pazopanib.
21. Pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2012-04; Primary Completion 2014-10 (Estimated); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | 30 months
  To asses the Objective Response (Complete Response or Partial Response) which provides second-line treatment with pazopanib in patients with carcinoma of advanced renal cell who have progressed or have not tolerated a first line of treatment with a Tyrosine Kinase Inhibitor.
  The Objective Response Rate will be evaluated using the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.

SECONDARY OUTCOMES:
Overall Survival | 30 months
  To assess the overall survival in patients treated with second-line treatment with pazopanib.
Treatment Safety Profile | 30 months
  To assess the treatment safety profile in patients treated with second-line treatment with pazopanib.
  Safety was assessed using Common Toxicity Criteria (CTC) of the National Cancer Institute (NCI), version 4.0.

CONTACTS AND LOCATIONS:
Overall Officials: Joaquim Bellmunt, MD, Study Chair — Hospital del Mar; Marta Guix, MD, Principal Investigator — Hospital del Mar; Juan Manuel Sepúlveda, MD, Principal Investigator — Hospital 12 de Octubre; Enrique Gallardo, MD, Principal Investigator — Corporació Sanitaria Parc Taulí; Xavier García del Muro, MD, Principal Investigator — Hospital Universitari de Bellvitge; Olatz Etxaniz, MD, Principal Investigator — Germans Trias i Pujol Hospital; José Luis González Larriba, MD, Principal Investigator — Hospital San Carlos, Madrid; Jose Angel Arranz, MD, Principal Investigator — Hospital General Universitario Gregorio Marañón; Emilio Esteban, MD, Principal Investigator — Hospital Universitario Central de Asturias; Aranzazu González del Alba, MD, Principal Investigator — Hospital Son Espases; Pablo Maroto, MD, Principal Investigator — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Locations (10):
- Spain (10):
  - Hospital Universitari Son Espases, Palma de Mallorca, Balearic Islands
  - Hospital Universitari Germans Trias i Pujol, Badalona, Barcelona
  - Hospital del Mar, Barcelona, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona, Barcelona
  - Hospital de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Corporació Sanitaria Parc Taulí, Sabadell, Barcelona
  - Hospital General Universitario Gregorio Marañón, Madrid, Madrid
  - Hospital 12 de Octubre, Madrid, Madrid
  - Hospital Clínico San Carlos, Madrid, Madrid
  - Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias